CLINICAL TRIAL: NCT06233513
Title: Behavioral and Neural Measures of Speech Motor Control
Brief Title: Vowel Space Expansion Sensorimotor Adaptation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017-1128 Adaptation (Exp 1-4); Protocol Version 10/31/2021 (Other: UW Madison); A481800 (Other: UW Madison); 1R01DC019134-01A1 (NIH)
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-08

CONDITIONS: Speech
Keywords: speech motor control; vocal learning
MeSH Terms: conditions — Speech

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Adult Speakers (Experimental): healthy adult participants across the lifespan in three groups:18-35, 36-55, and 56+
  Interventions: Behavioral: Exp 3 Speaking Task

INTERVENTIONS:
Behavioral: Exp 3 Speaking Task — Participant will sit in front of a computer screen in a quiet room and to produce speech based on what is on the screen. Participant may see real words or nonsense words to read. Investigators may play sounds through headphones and ask the participant to repeat them. Participant speech will be recorded by a microphone. This task takes about one hour to complete.
  Other Names: vowel space expansion

SUMMARY:
The purpose of this research study is to understand how the brain processes and controls speech in healthy people. The investigators are doing this research because it will help identify the mechanisms that allow people to perceive their own speech errors and to learn new speech sounds. 117 participants will be enrolled into this part of the study and can expect to be on study between 1 day (Experiment 1) and 4 weeks (Experiment 2).

DETAILED DESCRIPTION:
The overall study (Establishing the clinical utility of sensorimotor adaptation for speech rehabilitation) aims to understand how cognitive, perceptual, and motor processes are integrated in the control of speech movements. The investigators study how this complex skill is performed in healthy speakers to understand how this system functions, how this skill relates to the perception of speech, and what role different parts of the brain play in this process. Different studies look at how speech motor control is executed, maintained, and changed. Overall, the study will recruit 329 participants over the course of 5 years. Participants can expect to be on study for up to 4 weeks.

The entire study is composed of 8 experiments and 6 interventions. The present record represents Experiments 1-4: 1) Generalization of Vowel Space Expansion to Untrained Words and Vowels; 2) Retention of Vowel Space Expansion After Training in Multiple Sessions; 3) Vowel Space Expansion Training With Connected Speech, and 4)The Relationship Between Acuity, Variability, and Adaptation in Vowels. The paradigms in Experiments 1-3 all involve speech production under conditions of altered auditory feedback, while Experiment 4 is a correlative analysis that compares data from Experiments 1 and 2.

The Experiment 1 paradigm tests how the vowel space expansion induced by sensorimotor adaptation generalizes to untrained items in a single session. Participants will produce four training words (bead, bad, bod, and booed) under a vowel centralization feedback paradigm in which auditory feedback is altered, training them to produce these words with more vowel contrast. In addition to these trained words, eight test items will be produced in pre-training and post-training phases only. We will compare to measure how learning transfers across words that share the same vowel (test words: keep, cap, cop, coop) or whose vowels are intermediate to those of the trained words and which share consonants with the trained words (test words: bid, bud, bade, bode).

The Experiment 2 paradigm tests how the vowel space expansion induced by sensorimotor adaptation is retained over time. Participants will complete eight sessions of the vowel centralization sensorimotor adaptation paradigm over four weeks, producing four training words (bead, bad, bod, and booed) under conditions of altered auditory feedback that train them to produce these words with more vowel contrast. We will measure changes in produced vowels at the start of each session in a baseline phase to assess how much retained across days and weeks.

The Experiment 3 paradigm tests whether vowel space expansion can be evoked by a vowel centralization feedback paradigm applied to running speech (full sentences) rather than single words in healthy speakers. Participants will produce sentences from the Harvard corpus while their speech feedback is altered to centralize vowel feedback. The investigators will measure how working vowel space increases under this paradigm.

Experiment 4 is a correlative analysis which tests whether sensory acuity and speech production variability can predict magnitude of sensorimotor adaptation in interventions 1 and 2. Auditory acuity will be measured through a phoneme discrimination task in which vowel sounds are played to participants over headphones; somatosensory acuity will be measured through a tactile discrimination task in which participants report the orientation (horizontal or vertical) of the gratings on a plastic dome pressed lightly into the tongue. Speech production variability will be measured as the formant variability in the baseline phase of the sensorimotor adaptation experiments in interventions 1 and 2. These measures will be correlated with sensorimotor adaptation magnitude found in the prior interventions.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adults
* normal hearing and speech
* no history of stroke or neurological conditions

Exclusion Criteria:

* Native language other than English
* Any neurological disorders other than the disorder of interest
* Any history of hearing disorders
* Uncorrected vision problems that prevent participants from seeing visually-presented stimuli
* Significant cognitive impairments that prevent participants from carrying out the task or from giving informed consent
* Vulnerable populations (minors and prisoners)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Average Vowel Spacing (AVS) Measured as the Mean of Pairwise Formant Distances Between Vowels | up to 1 hour (Exp 1,3); eight visits of 1 hour each over 4 weeks (Exp 2)
  AVS is a local measure of vowel spacing.
Quadrilateral Vowel Space Area (qVSA) | up to 1 hour (Exp 1,3); eight visits of 1 hour each over 4 weeks (Exp 2)
  qVSA measures the area (in Hz^2) between the F1/F2 coordinates of the corner vowels. This is a global measure of working vowel space.
Intelligibility measured by Percent of words correctly identified by 5 independent transcribers | up to 1 hour (Exp 1,3); eight visits of 1 hour each over 4 weeks (Exp 2)
  Intelligibility is a perceptual measure. Four repetitions of each spoken production from each adaptation phase, as well as the minimal-pair neighbors from the calibration phase, will be identified by all transcribers. Because intelligibility in healthy speakers is expected to be near ceiling, speech signals will be masked by speech-shaped noise and delivered at 72 dB over closed-ear headphones. Signal-to-noise ratio will be determined prior to testing as the ratio where, on average, 50% of stimuli in the calibration phase are correctly identified. Transcribers will be native English speakers with no history of neurological/hearing disorders who pass a pure-tone hearing test.
Auditory acuity is measured as the average just noticeable difference (JND) along 4 vowel formant continua | up to 1 hour (Exp 1,3); eight visits of 1 hour each over 4 weeks (Exp 2)
  Auditory acuity is measured as the average just noticeable difference (JND) along 4 vowel formant continua: /i/-/ɪ/, /ɛ/-/æ/, /u/-/ʊ/, and /ɑ/-/ʌ/. Acuity will be measured at continua midpoint (across-category acuity) and at the four corner vowel endpoints (within-category acuity). JNDs will be measured through a 4-interval, 2-alternative forced choice task (AABA or ABAA) via a staircase procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Niziolek, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Link to study record for experiment 7 [NCT05723575] — https://clinicaltrials.gov/study/NCT05723575
- See also: Link to study record for experiment 5 [NCT05286658] — https://clinicaltrials.gov/study/NCT05286658